CLINICAL TRIAL: NCT06433921
Title: A Phase 1, Randomized, 2-part, 7-way Cross-over (Part 1) and 7-way Cross-over (Part 2), Blinded, Single Dose Study in Mild Asthmatics Aged 18-65 to Assess the Relative Potency of Salbutamol Administered Via Metered Dose Inhalers Containing Propellants HFA-152a (Test) and HFA-134a (Reference) Via Methacholine Bronchoprovocation and Systemic Pharmacodynamic Effects
Brief Title: A Study to Compare the Relative Potency of Salbutamol Administered Via Metered Dose Inhalers (MDI) Containing Propellants HFA-152a to HFA-134a in Mild Asthmatics Aged 18 to 65 Inclusive
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 219729; 2024-511220-14 (EudraCT Number)
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Asthma; Mild Asthma
Keywords: Salbutamol; Propellant HFA-152a; Propellant HFA-134a; Metered dose inhalers; Mild asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: 2-part, 7-way cross- over (Part 1 and Part 2)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Click here to enter text.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): Part 1 will consist of a 7 treatment, 7 period cross-over evaluation with all participants receiving the following treatments once, randomized to varying pre-specified sequences of:
  * Zero dose (placebo of both salbutamol HFA-134a and salbutamol HFA-152a)
  * 100 μg salbutamol HFA-134a
  * 200 μg salbutamol HFA-134a
  * 400 μg salbutamol HFA-134a
  * 100 μg salbutamol HFA-152a
  * 200 μg salbutamol HFA-152a
  * 400 μg salbutamol HFA-152a
  A minimum of a 2-day and maximum of a 7-day methacholine washout will separate each treatment period.
  Interventions: Drug: Salbutamol HFA-152a; Drug: Salbutamol HFA-134a; Drug: Placebo
- Part 2 (Experimental): Part 2 will consist of a 7 treatment, 7-way cross-over with all participants receiving the following treatments given once, randomized to varying pre-specified sequences of:
  * Zero dose (placebo of both salbutamol HFA-134a and salbutamol HFA-152a)
  * 100 μg salbutamol HFA-134a
  * 200 μg salbutamol HFA-134a
  * 400 μg salbutamol HFA-134a
  * 100 μg salbutamol HFA-152a
  * 200 μg salbutamol HFA-152a
  * 400 μg salbutamol HFA-152a
  A minimum of a 2-day and maximum of a 7-day methacholine washout will separate each treatment period.
  Interventions: Drug: Salbutamol HFA-152a; Drug: Salbutamol HFA-134a; Drug: Placebo

INTERVENTIONS:
Drug: Salbutamol HFA-152a — A single 100, 200 or 400 μg dose, given as 1, 2 or 4 × 100 μg actuations (exvalve) at 20 second intervals.
Drug: Salbutamol HFA-134a — A single 100, 200 or 400 μg dose, given as 1, 2 or 4 × 100 μg actuations (exvalve) at 20 second intervals.
Drug: Placebo — A single placebo HFA-152a suspension or placebo HFA-134a suspension dose, given as at 20 second intervals.

SUMMARY:
The primary objectives of the study are: Part 1: to characterize the potency and variability of dose response on efficacy (Provocative concentration of methacholine causing at least a 20% fall in forced expiratory volume (FEV1) [PC20]) of salbutamol administered via MDI with salbutamol HFA-134a or salbutamol HFA-152a in participants with mild asthma. Part 2: to compare the comparative dose response on efficacy (PC20) of salbutamol when administered via MDI with salbutamol HFA-134a or salbutamol HFA-152a in participants with mild asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; females may be of childbearing potential, of nonchildbearing potential, or postmenopausal.
2. Participant must be 18 to 65 years of age inclusive, at the time of screening.
3. ≥50 kg, at the time of screening.
4. Body mass index (BMI) with 19.0-35.0 kg/m2 inclusive, at the time of screening.

4. Documented history of asthma ≥ 6 months. 5. Receiving 1 of following asthma treatments, at a stable dose, for at least 12 weeks prior to the screening visit and is anticipated to remain stable for the duration of the study: i. Short-acting beta-agonist (SABA) only. ii. Daily maintenance low-dose inhaled corticosteroids (ICS) (defined as 100-250 μg/day fluticasone propionate or equivalent plus or minus SABA which is anticipated to remain stable for the duration of the study.

iii. Daily maintenance low-dose ICS + Long-acting beta-2 agonist (LABA) therapy (low-dose ICS defined as 100-250 μg/day fluticasone propionate or equivalent as defined by GINA [GINA, 2023]) plus or minus SABA, which is anticipated to remain stable for the duration of the study.

6. No severe asthma exacerbations within 6 months prior to screening and ≤1 severe exacerbation during the 12 months prior to screening.

7. Pre-bronchodilator FEV1 ≥80% of predicted, at screening. 8. PC20 to methacholine of ≤8 mg/mL, at screening. 9. Participants should be able to withhold SABA for ≥8 hours and LABA-containing medications for ≥48 hours for the purposes of performing the spirometry and methacholine challenge at screening and during the study visits (treatment periods).

10. A female participant is eligible to participate if she is not pregnant or breastfeeding, and Is a woman of woman of nonchildbearing potential (WONCBP) OR ii. Is a woman of child bearing potential (WOCBP) and using a contraceptive method that is highly effective.

11. Provide signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol.

12. Non-smokers who have not used any tobacco containing-products within 12 months prior to study start, and with a total pack year history of ≤10 pack years.

Exclusion Criteria:

1. Medical Conditions

   1. A history of life-threatening asthma or asthma that is unstable in the opinion of the investigator.
   2. A history of respiratory diseases to include (but not limited to): pneumothorax, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, cystic fibrosis, bronchiectasis, interstitial lung disease, emphysema, chronic obstructive pulmonary disease, tuberculosis, or other respiratory abnormalities other than asthma.
   3. Asymptomatic gallstones.
   4. History or current evidence of hematologic, neurologic, psychiatric, or other diseases that, in the opinion of the investigator, would put the participant at risk through study participation, or would affect the study analyses if the disease exacerbates during the study.
   5. Recent eye surgery or any other condition in which raised intracranial pressure (caused by forceful exhalation) would be harmful.
   6. Current use of cholinesterase inhibitor medication e.g., to treat myasthenia gravis.
2. Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day or participation in a clinical study within 30 days of study start, or 5 half-lives of study drug if that is longer.
3. Participants who are currently or in the last 15 days have worked nightshifts.
4. Regular alcohol consumption within 6 months prior to the study defined as: an average weekly intake of >21 units for males or >14 units for females.
5. A positive test result for drugs of abuse (including tetrahydrocannabinol) at screening or Day -1.
6. Use of combustible tobacco products, and non-combustible nicotine delivery systems, inclusive of cigarettes, cigars, pipes, and materials used to "vape" within 12 months prior to the start of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-06 (Estimated)

PRIMARY OUTCOMES:
Provocative concentration of methacholine causing at least a 20% fall in FEV1 (PC20) | Up to 11 weeks

SECONDARY OUTCOMES:
Peak QTc Interval | Up to 11 weeks
Peak Heart Rate (HR) | Up to 11 weeks
Minimum Serum Potassium | Up to 11 weeks
Maximum Observed Plasma Concentration (Cmax) | Up to 11 weeks
Time to Reach Cmax (Tmax) | Up to 11 weeks
Area Under the Plasma Concentration-time Curve up to Last Time With Concentrations Above the Lower Limit of Quantification (LLOQ) (AUC[0-last]) | Up to 11 weeks
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 11 weeks
Absolute Values for 12-lead Electrocardiogram (ECG) Recording of HR | Up to 11 weeks
Absolute Values for 12-lead ECGs Recording of Intervals | Up to 11 weeks
  Intervals recorded: - PR. - QRS. - QT. - QTc
Change from Baseline for Post-dose 12-lead ECGs Recording of HR | Baseline and up to 11 weeks
  The 3 predose measures will be recorded and will be averaged for HR to derive 1 baseline value.
Change from Baseline for Post-dose 12-lead ECGs Recording of Intervals | Up to 11 weeks
  The 3 predose measures will be recorded and will be averaged for QTc interval to derive 1 baseline value. Intervals recorded: - PR. - QRS. - QT. - QTc
Number of Participants with Clinically Significant Changes in Clinical Laboratory Parameters | Up to 11 weeks
Absolute Values of Vital Signs (Systolic and Diastolic Blood Pressure) | Up to 11 weeks
Absolute Values of Vital Signs (Pulse Rate) | Up to 11 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/